CLINICAL TRIAL: NCT04588363
Title: An Observational Cohort Study to Determine Late Outcomes and Immunological Responses After Infection With SARS-CoV-2 in Children With and Without Multisystem Inflammatory Syndrome (MIS-C)
Brief Title: COVID-19: Pediatric Research Immune Network on SARS-CoV-2 and MIS-C
Acronym: PRISM
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); Clinical Trials in Organ Transplantation in Children (Other)
Responsible Party: Sponsor
Other Study IDs: DAIT PRISM-01; NIAID CRMS ID#: 38772 (Other: DAIT NIAID)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2); Multisystem Inflammatory Syndrome in Children (MIS-C); Coronavirus Disease 2019 (COVID-19)
Keywords: participants <21 years of age; observational cohort study; immunological responses post infection
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Nasal Swabs, Saliva, Stools, Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SARS-CoV-2 positive children: Individuals less than 21 years of age who fulfill one or more of the following criteria:
  * SARS-CoV-2 detection from a respiratory specimen, and/or
  * Meets criteria for MIS-C, and/or
  * Meets criteria for MIS-C, except has involvement of only 1 organ system
  Interventions: Other: SARS-CoV-2 and/or MIS-C Exposure

INTERVENTIONS:
Other: SARS-CoV-2 and/or MIS-C Exposure — This is an observational cohort study.
  Other Names: Exposure: Severe Acute Respiratory Syndrome Coronavirus 2 Infection and/or Multisystem Inflammatory Syndrome in Children diagnosis

SUMMARY:
The primary objectives of this study are:

* To determine the proportion of children with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) related death, rehospitalization or major complications after infection with SARS-CoV-2 and/or Multisystem Inflammatory Syndrome in Children (MIS-C), and
* To determine immunologic mechanisms and immune signatures associated with disease spectrum and subsequent clinical course during the year of follow-up.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational cohort study to assess short and long-term clinical outcomes and immune responses after Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection and/or Multisystem Inflammatory Syndrome in Children (MIS-C) in children (e.g., defined as individuals who have not reached their 21st birthday at the time of enrollment). SARS-CoV-2 causes Coronavirus Disease 2019 (COVID-19)

Participants will be identified through active recruitment measures within hospitals and through ambulatory and laboratory-based databases of SARS-CoV-2 positive individuals <21 years of age. The study will enroll a minimum of 250 subjects from a diverse racial/ethnic background, from participating medical centers in the United States. The study period of participation is 1 year (12 months).

ELIGIBILITY:
Inclusion Criteria:

1. Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) detection from a respiratory specimen, and/or
2. Meets criteria for Multisystem Inflammatory Syndrome in Children (MIS-C), and/or
3. Meets criteria for MIS-C, except has involvement of only 1 organ system

Cases meeting clinical criteria for MIS-C but without known SARS-CoV-2 exposure, and who are being treated as MIS-C by the treating physician, but with negative SARS-CoV-2 PCR and pending or negative antibody testing, may be enrolled as subjects. If subsequent antibody testing is positive, cases will be labelled as confirmed MIS-C. If SARS-CoV-2 antibody testing is negative, subjects will be labeled at the end of the study as suspected/not confirmed MIS-C.

Exclusion Criteria:

1. Subject and/or parent/guardian who are not able to understand or be willing to provide informed consent and where applicable assent

--Note, for this observational cohort study, participation in other COVID-19 studies is not an automatic exclusionary criterion.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Individuals less than 21 years of age who fulfill one or more of the following criteria:
  * SARS-CoV-2 detection from a respiratory specimen, and/or
  * Meets criteria for MIS-C, and/or
  * Meets criteria for MIS-C, except has involvement of only 1 organ system
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Either COVID-19-Related Death, Rehospitalization, Major Complications after SARS-CoV-2 Illness and/or MIS-C at 6 Months Post Illness Presentation | 6 Months Post Illness Presentation (Enrollment)
  Participants who experience Coronavirus Disease 2019 (COVID-19)-related death, rehospitalization or major complications after Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) illness and/or multisystem inflammatory syndrome in children (MIS-C).

SECONDARY OUTCOMES:
Proportion of Participants with Coronavirus Disease 2019 (COVID-19)-Related Death after Multisystem Inflammatory Syndrome in Children (MIS-C) at 1 Year Post Illness Presentation | 1 Year Post Illness Presentation (Enrollment)
  Participants who experience Coronavirus Disease 2019 (COVID-19)-related death, rehospitalization or major complications after Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) illness and/or multisystem inflammatory syndrome in children (MIS-C).
All-Cause Mortality | 1 Year Post Illness Presentation (Enrollment)
  The occurrence of death in participants regardless of relationship to Coronavirus Disease 2019 (COVID-19) and Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2).
Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Mortality | 1 Year Post Illness Presentation (Enrollment)
  The occurrence of SARS-CoV-2 related death in participants.
Hospitalization for Participants Enrolled as an Outpatient or Rehospitalization after First Admission in Hospitalized Participants | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of Participants who require:
  * Hospitalization subsequent to enrollment as an outpatient for SARS-CoV-2/COVID-19 related illness and/or MIS-C, or
  * Rehospitalization after discharge from their initial admission for SARS-CoV-2/COVID-19 related illness and/or MIS-C.
  Abbreviations:
  * Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
  * Coronavirus Disease 2019 (COVID-19)
  * Multisystem Inflammatory Syndrome in Children (MIS-C)
Coagulation Abnormality by D-Dimer Biomarker | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of dysregulation involving the coagulation system by D-dimer laboratory test.
Coagulation Abnormality by Fibrinogen Biomarker | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of dysregulation involving the coagulation system by fibrinogen laboratory test.
Coagulation Abnormality by Prothrombin Time (PT) and Activated Partial Thromboplastin Time (PTT) Biomarkers | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of dysregulation involving the coagulation system by PT and PTT laboratory tests.
Coagulation Abnormality by International Normalised Ratio (INR) Biomarker | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of dysregulation involving the coagulation system by INR laboratory test.
Coronary Artery Abnormalities | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of coronary artery abnormalities (e.g., by echocardiogram and, if performed for clinical indications, angiogram, as examples).
Pulmonary Hypertension | Up to 1 Year Post Illness Presentation (Enrollment)
  Prevalence of pulmonary hypertension by echocardiogram and standard of care assessments.
Cardiovascular System Dysregulation by B-type natriuretic peptide (BNP) Biomarker | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of cardiovascular system dysregulation by BNP laboratory test.
Cardiovascular System Dysregulation by Troponin I Biomarker | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of cardiovascular system dysregulation by Troponin I laboratory test.
Cardiovascular System Dysregulation by Echocardiogram | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of cardiac function by echocardiogram (Echo), a test that uses high frequency sound waves (ultrasound) to make pictures of the heart. The test is also referred to as a diagnostic cardiac ultrasound.
Cardiovascular System Dysregulation by Electrocardiogram (ECG) | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of cardiovascular system dysregulation(s) evaluated by standardized 12-lead electrocardiogram. ECG rhythms, intervals and voltages will be assessed. Cross reference: ECG and EKG are used interchangeably.
Pulmonary Abnormalities | Up to 1 Year Post Illness Presentation (Enrollment)
  Pulmonary fibrosis (i.e., scarring) or other abnormalities detected by computerized tomography (CT) imaging.
Pulmonary Function Characteristics | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization by pulmonary function tests (spirometry without bronchodilators).
Renal/Metabolic Biomarkers: Serum Creatinine and Blood Urea Nitrogen (BUN) | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of kidney/metabolic function by serum creatinine and blood urea nitrogen (BUN) laboratory tests
Renal/Metabolic Biomarker: Estimated glomerular filtration rate (eGFR) | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of kidney/metabolic function by the estimated glomerular filtration rate (eGFR) calculated value, using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
Hepatic/Metabolic Biomarkers: Serum Alkaline Phosphatase (Alk Phos), Alanine Aminotransferase ( ALT/SGPT)and Aspartate Aminotransferase (AST/SGOT) | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of liver/metabolic function by the following laboratory tests:
  * alkaline phosphatase
  * alanine aminotransferase (ALT/SGPT) and
  * aspartate aminotransferase (AST/SGOT).
Hepatic/Metabolic Biomarker: Total Bilirubin | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of liver/metabolic function by serum total bilirubin laboratory test.
Neurologic Abnormalities | Up to 1 Year Post Illness Presentation (Enrollment)
  Characterization of neurologic sequelae of infection/disease.
Other End Organ and/or functional abnormalities Occurring After Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection/ Coronavirus Disease 2019 (COVID-19) and/or Multisystem Inflammatory Syndrome in Children (MIS-C) | Up to 1 Year Post Illness Presentation (Enrollment)
  Identified by and characterized during standard of care assessments.
Health Related Quality of Life | Up to 1 Year Post Illness Presentation (Enrollment)
  Assessment of health-related quality of life (HRQOL) after Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection/ Coronavirus Disease 2019 (COVID-19) and/or multisystem inflammatory syndrome in children (MIS-C).
  The Pediatric Quality of Life Inventory is a series of assessment instruments designed to measure the health-related quality of life of children. The PedsQL 4.0 provides an opportunity for the assessment of both overall (generic) quality of life as well as disease-specific quality of life.
  The PedsQL 4.0 Generic Core Scales are appropriate for assessing health-related quality of life in both healthy and chronically ill children. The four scales making up this generic battery include Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items).

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Webber, MBChB, MRCP, Study Chair — Department of Pediatrics, Monroe Carell Jr. Children's Hospital at Vanderbilt; James D. Wilkinson, MD, MPH, Principal Investigator — Vanderbilt Institute for Clinical and Translational Research (VICTR); Natasha B Halasa, MD, MPH, Principal Investigator — Department of Pediatrics, Vanderbilt University Medical Center; Virginia Pascual, MD, Principal Investigator — Gale and Ira Drukier Institute for Children's Health, Weill Cornell Medicine; Betty Diamond, MD, Principal Investigator — Institute of Molecular Medicine, The Feinstein Institute for Medical Research; Ignacio Sanz, MD, Principal Investigator — Division of Rheumatology, Emory University; Olivia Martinez, PhD, Principal Investigator — Stanford University; Sheri Krams, PhD, Principal Investigator — Stanford University; Jeremy Boss, PhD, Principal Investigator — Emory University
Locations (20):
- United States (20):
  - Loma Linda University Health, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Mayo Clinic Rochester, Rochester, Minnesota
  - St. Louis Children's Hospital, St Louis, Missouri
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - NewYork-Presbyterian Queens Hospital, Flushing, New York
  - Cohen Children's Medical Center - Northwell Health, New Hyde Park, New York
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - NewYork-Presbyterian Komansky Children's Hospital, New York, New York
  - Mount Sinai Kravis Children's Hospital, New York, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Duke University Children's Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Pediatric Rheumatology, Charleston, South Carolina
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee

REFERENCES:
- See also: Clinical Trials in Organ Transplantation in Children — https://www.ctotc.org/
- See also: Division of Allergy, Immunology and Transplantation — http://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infection Diseases — https://www.niaid.nih.gov/